CLINICAL TRIAL: NCT07228169
Title: Feasibility and Effectiveness of a Multimodal Exercise Intervention on Physical Activity and Physical Functions in Low-Income Older Adults
Brief Title: Tai Chi Interventions on Physical Functions Among Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Weiyun Chen, Associate Professor, University of Michigan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: HUM00267001
Record Dates: First submitted 2025-10-19; First posted 2025-11-14 (Actual); Last update posted 2025-11-14 (Actual); Status verified 2025-11

CONDITIONS: Combined Multicomponent Exercise and Tai Chi
Keywords: Multicomponent exercise; Tai Chi; Physical activity; Physical function
MeSH Terms: conditions — Motor Activity | interventions — Tai Ji

STUDY DESIGN:
Intervention Model Description: Participants attended one 45-minute multicomponent exercise group session and one 45-minute Tai Chi group session each week for eights weeks, along with self-practice.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Combined multicomponent exercise and Tai Chi (Experimental): This combined multicomponent exercise and Tai Chi intervention includes that participants attended one 45-minute multicomponent exercise group session and one 45-minute Tai Chi group session each week, along with self-practice for eight weeks.
  Interventions: Behavioral: Combined multicomponent exercise and Tai Chi

INTERVENTIONS:
Behavioral: Combined multicomponent exercise and Tai Chi — The combined multicomponent exercise and Tai Chi intervention includes that participants attended one 45-minute multicomponent exercise group session and one 45-minute Tai Chi group sessions along with self-practice each week, for eight weeks.

SUMMARY:
This study examined the feasibility and effectiveness of a multimodal exercise intervention on an objective measure of physical activity (PA), and objective and subjective measures of physical functions among older adults living in a low-income senior housing complex.

DETAILED DESCRIPTION:
This study aimed to examine the feasibility and effectiveness of a multimodal exercise intervention on an objective measure of physical activity (PA), and objective and subjective measures of physical functions among older adults living in a low-income senior housing complex. 23 older adults (mean age = 80.17 ± 6.913 years) residing in a low-income senior housing complex voluntarily participated in an 8-week intervention. The feasibility of the study was assessed throughout the study period. Additionally, participants completed The Acceptability, Appropriateness, and Feasibility of the Intervention Questionnaire (AAF-IQ) after the intervention. The study outcomes, including physical activity and physical functions, were measured within two weeks before and after the intervention.

ELIGIBILITY:
Inclusion Criteria:

1. age 65 years or above,
2. able to walk for 10 feet without human assistance, a cane or walker was permitted,
3. willing to wear an ActiGraph activity monitor for 7 days at baseline and post-intervention test,
4. exercise safely as determined by their healthcare provider,
5. complete the study tests and questionnaires,
6. sign the informed consent,
7. able and willing to comply with the requirements of the protocol.

Exclusion Criteria:

1. having recent medical limitations including recent myocardial infarction, stroke, or physical limitations for exercises by completing the Physical Activity Readiness Questionnaire (PAR-Q),
2. having 40 or higher body mass index (BMI) by self-reporting body weight and body height, inputting these into the computerized BMI calculator.

Ages: 65 Years to 95 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Gender Based: Yes — males and females.
Enrollment: 27 (Actual)
Dates: Start 2025-02-27 (Actual); Primary Completion 2025-05-14 (Actual); Study Completion 2025-09-23 (Actual)

PRIMARY OUTCOMES:
Weekly Physical Activity Minutes | Baseline test and post-intervention test (up to 3 months).
  Weekly physical activity minutes were measured by having participants wear an ActiGraph activity monitor for seven consecutive days during waking hours, expect for bathing activities. The raw data were analyzed by using the ActiLife software.
Short Physical Performance Battery (SPPB)-Repeated Chair Stand test. | Baseline test and post-intervention test (up to 3 months).
  This test is used to measure low extremity strength.
The Short Physical Performance Battery-Balance test. | Baseline and post-intervention test (Up to 3 months).
  This test is used to measure balance.

SECONDARY OUTCOMES:
Timed Up and Go Test | Baseline test and the post-intervention test (up to 3 months).
  This test is used to measure gait speed.
The Patient-Reported Outcomes Measurement Information System (PROMIS) Physical Function Short Form | Baseline test and post-intervention test (up to 3 months).
  This questionnaire is used to assess participants' perceived physical function.
Assessing Feasibility, Acceptability, and Appropriateness of the Intervention Questionnaire | Post-intervention test (up to one week).
  This questionnaire is used to assess the participant's views of feasibility, acceptability, and appropriateness of the intervention.

CONTACTS AND LOCATIONS:
Locations (1):
- School of Kinesiology, University of Michigan, Ann Arbor, Michigan, United States